CLINICAL TRIAL: NCT00788710
Title: A Double-Blind, Placebo-Controlled, Multicenter Trial to Study the Efficacy and Tolerability of MK0663/Etoricoxib in the Treatment of Pain After Abdominal Hysterectomy
Brief Title: A Study of MK0663/Etoricoxib for Post-Abdominal Hysterectomy Surgery Pain (0663-097)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-097; 2008_578
Record Dates: First submitted 2008-11-05; First posted 2008-11-11 (Estimated); Results first posted 2011-07-22 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Acute Pain Following a Total Abdominal Hysterectomy
MeSH Terms: interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Etoricoxib 120 mg (Experimental): etoricoxib (MK0663) 120 mg (2 60 mg tablets) and 1 placebo tablet once daily on Days 1-5. Total treatment is 5 days.
  Interventions: Drug: etoricoxib (MK0663) 120 mg
- Etoricoxib 90 mg (Experimental): etoricoxib (MK0663) 90 mg tablet and 2 placebo tablets once daily on Days 1-5. Total treatment is 5 days.
  Interventions: Drug: etoricoxib (MK0663) 90 mg
- Placebo (Placebo Comparator): Placebo- 3 tablets once daily
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: etoricoxib (MK0663) 120 mg — 120 mg of etoricoxib (MK0663) for a total of 5 days
  Other Names: Arcoxia
  Arms: Etoricoxib 120 mg
Drug: Comparator: Placebo — Placebo tablets once daily on Days 1-5. Total treatment is 5 days.
  Arms: Placebo
Drug: etoricoxib (MK0663) 90 mg — 90 mg of etoricoxib (MK0663) for a total of 5 days
  Arms: Etoricoxib 90 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of etoricoxib compared to placebo in the treatment of postoperative pain associated with total abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older in generally good health who are scheduled to have a total hysterectomy and who are willing to limit alcohol consumption

Exclusion Criteria:

* Patient is allergic to the study drug, other cyclooxygenase-2 (COX-2) inhibitors/nonsteroidal anti-inflammatory drugs (NSAIDS), ibuprofen, morphine, or oxycodone or has hypersensitivity to aspirin or other NSAIDS
* Patient has uncontrolled high blood pressure
* Patient has a history of drug and/or alcohol abuse within the last 5 years
* Patient has taken part in another investigational study within 4 weeks of the start of study
* Patient is breast-feeding
* Patient has an active ulcer or inflammatory bowel disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Viscusi ER, Frenkl TL, Hartrick CT, Rawal N, Kehlet H, Papanicolaou D, Gammaitoni A, Ko AT, Morgan LM, Mehta A, Curtis SP, Peloso PM. Perioperative use of etoricoxib reduces pain and opioid side-effects after total abdominal hysterectomy: a double-blind, randomized, placebo-controlled phase III study. Curr Med Res Opin. 2012 Aug;28(8):1323-35. doi: 10.1185/03007995.2012.707121. Epub 2012 Jul 16. PMID 22738802

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo - 3 tablets once daily on Days 1-5. Total treatment is 5 days.
Period: Overall Study
Arm/Group | Etoricoxib 120 mg | Etoricoxib 90 mg | Placebo
Started | 144 | 142 | 144
Completed | 139 | 134 | 138
Not Completed | 5 | 8 | 6
Not completed — Adverse Event | 1 | 3 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etoricoxib 120 mg | Etoricoxib 90 mg | Placebo | Total
Number analyzed (Participants) | 144 | 142 | 144 | 430
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (6.9) | 47.0 (7.2) | 45.7 (7.0) | 46.3 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 142 | 144 | 430
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Intensity at Rest Over Days 1 to 3
Description: Pain intensity at rest was measured on a 0- to 10-point scale: 0=no pain, to 10=pain as bad as you can imagine.
Time Frame: 3 Days
Population: Full analysis set population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Etoricoxib 120 mg | Etoricoxib 90 mg | Placebo
Number analyzed (Participants) | 133 | 127 | 135
Score on a scale | 2.40 (0.15) | 2.46 (0.15) | 3.26 (0.15)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

2. Secondary Outcome: Average Total Daily Dose of Morphine Over Days 1 to 3
Time Frame: 3 days
Population: Full analysis set population
Measure: Least Squares Mean (Standard Error); unit: milligrams (mg)
Arm/Group | Etoricoxib 120 mg | Etoricoxib 90 mg | Placebo
Number analyzed (Participants) | 132 | 130 | 134
milligrams (mg) | 5.37 (0.08) | 5.46 (0.08) | 7.75 (0.08)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

3. Secondary Outcome: Average Elicited Pain Upon Sitting Over Days 1 to 3
Description: Elicited pain upon sitting was measured on a 0- to 10-point scale: 0=no pain, to 10=pain as bad as you can imagine.
Time Frame: 3 days
Population: Full analysis set population
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Etoricoxib 120 mg | Etoricoxib 90 mg | Placebo
Number analyzed (Participants) | 133 | 127 | 135
Score on a scale | 3.58 (0.17) | 3.80 (0.17) | 4.71 (0.17)
Statistical Analysis 1: Comparison: Etoricoxib 120 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Etoricoxib 90 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA

ADVERSE EVENTS:
Arm/Group | Etoricoxib 120 mg | Etoricoxib 90 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 5/144 | 5/142 | 10/144
Other Adverse Events (participants affected / at risk) | 60/144 | 51/142 | 65/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib 120 mg (N=144) | Etoricoxib 90 mg (N=142) | Placebo (N=144)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoricoxib 120 mg (N=144) | Etoricoxib 90 mg (N=142) | Placebo (N=144)
Constipation (Gastrointestinal disorders) | 16 (17) | 12 (13) | 18 (20)
Flatulence (Gastrointestinal disorders) | 7 (7) | 14 (14) | 12 (12)
Nausea (Gastrointestinal disorders) | 40 (41) | 31 (35) | 38 (43)
Vomiting (Gastrointestinal disorders) | 10 (10) | 7 (7) | 10 (10)
Pyrexia (General disorders) | 7 (7) | 4 (4) | 24 (27)
Dizziness (Nervous system disorders) | 12 (12) | 9 (9) | 14 (14)
Headache (Nervous system disorders) | 9 (11) | 8 (8) | 14 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 13 (14) | 6 (6)

LIMITATIONS AND CAVEATS:
11 participants were screened & 10 participants were randomized at site 0028. An audit showed study medication dispensing logs were not kept. These 10 participants were invalidated and excluded from both efficacy & safety analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.